CLINICAL TRIAL: NCT04789538
Title: Retro-prospective Evaluation of the Clinical Safety and Effectiveness of Hydrophilic Acrylic Intraocular Lens (509)
Brief Title: Safety and Effectiveness of an Hydrophilic Acrylic Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Other Study IDs: ASPHINA 509 BER-401-20
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2021-05

CONDITIONS: Cataract Senile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monofocal IOL
  Interventions: Other: monofocal lens

INTERVENTIONS:
Other: monofocal lens — not applicable as patients are already implanted with the monofocal intraocular lens

SUMMARY:
Evaluation of the clinical safety and effectiveness of hydrophilic acrylic intraocular lens

DETAILED DESCRIPTION:
To show safety and the effectiveness in regard to the monocular corrected distance visual acuity (CDVA) at 12-24 month postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any gender, aged 18 years or older at the time of the surgery
* Patients who had an uncomplicated (no intra-operative complication) aged-related cataract surgery
* Currently implanted with the study device into the capsular bag in at least one eye
* One-year post surgery follow-up (365 days -14 days/+365 days) for the study eye at the time of the postoperative visit
* Patient is willing and capable of providing informed consent
* Patient is willing and capable of complying with visits and procedures as defined by this protocol

Exclusion Criteria:

* Preoperative corrected distance visual acuity (CDVA) better than 0.3 LogMAR (0.5 decimal) or CDVA not available preoperatively
* Preoperative documented endothelial cell count of less than 2000/mm2 (if available)
* Any preoperative documented ocular disorder that could potentially cause a clinically significant future visual acuity loss
* Any preoperative documented clinically significant anterior segment pathology (e.g. chronic uveitis, iritis, aniridia, rubeosis iridis, anterior membrane dystrophies, poor pupil dilation, etc.)
* Any preoperative documented clinically significant abnormal corneal finding (e.g. keratoconus, pellucid marginal degeneration, or irregular astigmatism, clinically significant corneal membrane dystrophies)
* Any preoperative documented clinically significant condition that could affect IOL stability (e.g. zonular dialysis, evident zonular weakness or dehiscence, etc.)
* Any preoperative documented history of clinically significant retinal pathologies or ocular diagnosis (e.g. diabetic retinopathy, ischemic diseases, macular degeneration, retinal detachment, optic neuropathy optic nerve atrophy, amblyopia, strabismus, microphthalmos, aniridia, epiretinal membrane etc.) that could alter or limit final postoperative visual prognosis
* Any preoperative acute infection (acute ocular disease, external/internal infection, systemic infection)
* Any previous preoperative intraocular and corneal surgery
* Preoperative documented uncontrolled glaucoma or IOP higher than 24mmHg under ocular hypertension treatment
* Preoperative documented or current systemic or ocular pharmacotherapy that effects patients' vision
* Any other preoperative documented or current pathology or condition that could be a risk for the patient according to the investigator opinion
* Women during pregnancy and/or lactation at time of enrollment into the study
* Patients unable to meet the limitations of the protocol or likely of non-cooperation during the trial
* Patients whose freedom is impaired by administrative or legal order
* Subject is enrolled in any other concurrent clinical study, with the exception of local mandatory governmental registries and observational studies/registries, that do not affect patients' vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with the study lens IOLs
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 12 to 24 months after the implantation
  Visual acuity at far distance

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Desgenettes, Lyon, France